CLINICAL TRIAL: NCT01889563
Title: Potential Effects of 6 vs 12-weeks of Physical Training on Cardiac Autonomic Function and Functional Capacity in COPD
Brief Title: Physical Training and Heart Rate Variability in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Renata Goncalves Mendes, PhD, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: COPD6VS12
Record Dates: First submitted 2013-06-25; First posted 2013-06-28 (Estimated); Results first posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: chronic obstructive pulmonary disease; heart rate variability; physical training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical exercise training program (Experimental): Physical Exercise Training Program Exercise training was conducted in three times a week, during 12 weeks at high-intensity targets. Each session consisted of a five minute warm up (walking) at 2 km/h and 30 minutes with an intensity targets set at 70% of the peak speed rate. The increase of intensity was 0.5Km/h when the patient scored less than 4 point of Borg scale (moderate to intense effort) during each session. All evaluations were done at 6th week, in order to analyze the progression of outcomes and exactly adjust the intensity of training.
  Interventions: Other: Physical Exercise Training Program Exercise
- No Physical Exercise Training Program (No Intervention): No Physical Exercise Training Program

INTERVENTIONS:
Other: Physical Exercise Training Program Exercise — Physical Exercise Training Program Exercise training was conducted in three times a week, during 12 weeks at high-intensity targets. Each session consisted of a five minute warm up (walking) at 2 km/h and 30 minutes with an intensity targets set at 70% of the peak speed rate. The increase of intensity was 0.5Km/h when the patient scored less than 4 point of Borg scale (moderate to intense effort) during each session. All evaluations were done at 6th week, in order to analyze the progression of outcomes and exactly adjust the intensity of training.
  Arms: Physical exercise training program

SUMMARY:
To contrast the potential effects of physical exercise training program (PTP) of a 6 versus 12 weeks on cardiac autonomic modulation by linear and non-linear heart rate variability (HRV) indices and functional capacity in moderate-to-severe COPD patients.

DETAILED DESCRIPTION:
This is a prospective randomized controled trial. A total of fifty two patients were recruited, however, only 32 patients met all inclusion criteria. Patients that were included presented: 1) a diagnosis of COPD according to criteria set forth by the Global Initiative for Chronic Obstructive Lung Disease (19), 2) compliance with medical management, 3) no change in medical management and no decompensation episodes for at least one month prior to study initiation, and 4) no participation in a regular physical exercise program for at least six months prior to study initiation. Exclusion criteria consisted of the presence of orthopedic or neurological conditions that would preclude participation in a physical exercise program, a history of cardiac arrhythmias, a past history consistent with heart disease, diabetes mellitus, arterial hypertension and failure to comply with the research protocol.

Patients were randomly assigned to physical exercise training program PTG, (n=17) or to a control group (CG, n=15) without aerobic exercise training by drawing of shuffled, opaque, coded envelopes that were opened immediately before starting each case. However, after the randomization process, five patients refused to continue and seven interested patients were excluded.

Finally the groups were composed of PTG (n=10) and control group (CG, n=10). Heart rate variability (HRV) on rest and during submaximal test was determined by linear analysis (rMSSD and SDNN) and nonlinear indices SD1, SD2 and sample entropy (SE). In addition, the physiological responses were obtained during cardiopulmonary exercise testing (CPX), the walking distance (WD) on six minute walking test and submaximal constant speed testing (CST). PTP consisted of 30 minutes of aerobic exercise training on a treadmill, 3 times per week at 70% of CPX peak speed rate. Patients were evaluated on baseline, 6 and 12 weeks.

All patients received regular treatment consisting of inhaled bronchodilators and steroids and the dosage did not changed during the study. The study protocol was approved by the Institutional Ethics Committee and all patients signed a written consent form prior to study initiation (109/2006). The target number of patients was calculated to be 10 patients in each group, based on a 5% type I error, a 2-sided test, and an 80% power to detect a change between the groups in 5 to SD2 at rest. Considering a drop out of 20%, 12 patients in each group were calculated. Due to the Gaussian distribution and/or homogeneity of variance in variable values, parametric tests were selected for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of COPD according to criteria set forth by the Global Initiative for Chronic Obstructive Lung Disease (19),
2. compliance with medical management,
3. no change in medical management and no decompensation episodes for at least one month prior to study initiation, and
4. no participation in a regular physical exercise program for at least six months prior to study initiation.

Exclusion Criteria:

1. presence of orthopedic or neurological conditions that would preclude participation in a physical exercise program,
2. a history of cardiac arrhythmias,
3. a past history consistent with heart disease, diabetes mellitus, arterial hypertension and failure to comply with the research protocol.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-05; Primary Completion 2008-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Borghi-Silva, PhD, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Federal university f Sao Carlos, São Carlos, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Physical Exercise Training Program | No Physical Exercise Training Program
Started | 17 | 15
Completed | 10 | 10
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Exercise Training Program | No Physical Exercise Training Program | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (7) | 66 (10) | 66 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 14 | 10 | 24
Region of Enrollment [Number; unit: participants]
  Brazil | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: The SD1 Index, a Nonlinear Index of Heart Rate Variability (HRV)That Represents the Parassimpatetic Activity.
Description: Patients underwent the assessments proposed in the study on an outpatient basis before and after 6 and 12 weeks of physical exercise training program. The primary end-point measure was the SD1, a nonlinear index of HRV that represent the parasympathetic modulation
Time Frame: baseline (before physical exercise training program), 6 and 12 weeks after intervention
Measure: Mean (Standard Deviation); unit: miliseconds
Arm/Group | Physical Exercise Training Program | No Physical Exercise Training Program
Number analyzed (Participants) | 10 | 10
miliseconds
  Baseline | 3.7 (1.7) | 2.8 (1.4)
  After 6-weeks | 7.1 (3.6) | 2.5 (0.8)
  After 12-weeks | 13.6 (8.8) | 2.5 (1.3)

2. Secondary Outcome: Walking Distance on Six Minute Walking Test
Description: Patients underwent the assessments proposed in the study on an outpatient basis before physical exercise training program and after 6 and 12 weeks of physical exercise training program. The second end-point was walking distance on six minute walking test.
Time Frame: Baseline (before physical exercise training program) and after 6 and 12 weeks of physical exercise training program
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Physical Exercise Training Program | No Physical Exercise Training Program
Number analyzed (Participants) | 10 | 10
meters
  Baseline | 341 (210) | 327 (157)
  After 6-weeks | 596 (246) | 430 (159)
  After 12-weeks | 602 (307) | 424 (173)

ADVERSE EVENTS:
Arm/Group | Physical Exercise Training Program | No Physical Exercise Training Program
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 0/17 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No